CLINICAL TRIAL: NCT03425045
Title: Repetitive Transcranial Magnetic Stimulation for Chronic Subjective Non-Pulsatile Primary Tinnitus Compared to Placebo and Medicament Therapy
Brief Title: Repetitive Transcranial Magnetic Stimulation for Chronic Subjective Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FNO-ENT-tinnitus; MH CZ-DRO (FNOs/2015) (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2018-01-15; First posted 2018-02-07 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Tinnitus, Subjective
Keywords: chronic tinnitus; repetitive transcranial magnetic stimulation; hypacusion; depression; treatment; placebo; medication therapy
MeSH Terms: conditions — Tinnitus; Depression | interventions — Transcranial Magnetic Stimulation; Ginkgo biloba extract

STUDY DESIGN:
Intervention Model Description: The study is designed as interventional, blinded, randomized, controlled trial with three parallel arms
Who Masked: Participant, Outcomes Assessor
Masking Description: The study subjects and outcomes assessors will be masked, the investigator will know which treatment is being provided for which patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repetitive Transcranial Magnetic Stimulation (Experimental): Patients in this study arm will undergo the rTMS stimulation as described above.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation
- Sham stimulation (Sham Comparator): Patients in this study arm will undergo the sham stimulation as described above.
  Interventions: Procedure: Sham stimulation
- Ginkgo Biloba Extract (Active Comparator): Patients in this study arm will receive medication therapy as described above, without any rTMS or sham procedure.
  Interventions: Drug: Ginkgo Biloba Extract

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation — Patients randomised in Arm 1 will receive stimulation of the dorsolateral prefrontal cortex (frequency 25 Hz; 300 pulses; 80% resting motor threshold=RMT) and primary auditory cortex on both sides (1 Hz; 1000 pulses; 110% RMT) will be stimulated in patients in rTMS stimulation group for 5 consecutive days. No medication therapy will be provided for patients in this arm.
  Arms: Repetitive Transcranial Magnetic Stimulation
Procedure: Sham stimulation — Sham stimulation will be performed in patients randomised in Arm 2 of the study for 5 consecutive days. No medication therapy will be provided for patients in this arm.
  Arms: Sham stimulation
Drug: Ginkgo Biloba Extract — Patients randomised in Arm 3 of the study will receive medication therapy with Ginkgo biloba extract EGb 761 once a day for 6 months.
  Arms: Ginkgo Biloba Extract

SUMMARY:
Therapy of subjective chronic primary tinnitus could be challenging. Repetitive transcranial magnetic stimulation (rTMS) is currently being tested for suppressing the symptoms. However, effect of stimulation remains controversial. The aim was to uncover real effect of rTMS stimulation for tinnitus treatment. There will be three groups, stimulation group, sham stimulation group and controlled group with medicament treatment. The investigators assume that combination of rTMS stimulation of dorsolateral prefrontal cortex and primary auditory cortex at both sides will be more efficient. The investigators considered a 10% improvement in the tinnitus questionnaire score and in the tinnitus masking to be clinically relevant.

DETAILED DESCRIPTION:
Adult patients suffering from chronic subjective non-pulsatile primary unilateral or bilateral tinnitus for at least 6 months will be included in the study. Patients will be randomly assigned using a random number generation randomization method into rTMS stimulation group (group 1), sham stimulation group (group 2) and group with medicament therapy only (group 3). Dorsolateral prefrontal cortex (frequency 25 Hz; 300 pulses; 80% resting motor threshold=RMT) and primary auditory cortex on both sides (1 Hz; 1000 pulses; 110% RMT) will be stimulated in patients in rTMS stimulation group for 5 consecutive days. Both the patients and outcome assessor were blinded to the intervention group in which the patients (rTMS and shame stimulation group) belonged to. Medicament therapy in group 3 will consist of ginkgo biloba extract EGb 761 once a day for 6 months. There will be no medicament therapy for tinnitus in group 1 and 2. Tinnitus reaction questionnaire (TRQ), tinnitus handicap questionnaire (THQ), tinnitus handicap inventory (THI), Beck Depression Inventory (BDI), pure-tone audiometry with Fowler scoring of hearing loss and tinnitus analysis will be used for evaluation of tinnitus in all patients. Data will be recorded on the day patient is included in the study, during follow-up after 1 month and 6 months. Descriptive statistics, such as the arithmetic mean, standard deviation, and absolute and relative frequency tables, will be used for data processing. The Pearson's chi-squared test, Fisher's exact test, Kruskal-Wallis test and analysis of variance will be used for comparison. The statistical tests will be assessed using a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

- subjective chronic non-pulsatile tinnitus lasting more than 6 months

Exclusion Criteria:

* head injury or brain surgery
* epilepsy
* organic brain lesion
* Meniere's disease or fluctuating hearing loss
* cochlear or bone-anchored hearing device implantation
* history of suicide
* pregnancy
* therapy with anticonvulsants
* antipsychotic medication
* heart pacemaker implantation
* rTMS performed in the past
* not signing of the informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Tinnitus Reaction Questionnaire (TRQ) | 36 months
  This questionnaire will be used to find out what sort of effects tinnitus has had on the lifestyle and general well-being of the patients. 10% improvement will be considered clinically relevant.
Tinnitus Handicap Questionnaire (THQ) | 36 months
  This questionnaire has 27 questions and will be used to assess the degree of handicap that the tinnitus presents for the affected patients. 10% improvement will be considered clinically relevant.
Tinnitus Handicap Inventory (THI) | 36 months
  The purpose of this questionnaire is to identify difficulties the affected patients may be experiencing because of tinnitus. 10% improvement of the score will be considered clinically relevant.

SECONDARY OUTCOMES:
Improvement of depression - Beck Depression Inventory | 36 months
  Improvement of depressive symptoms in patients will be assessed using the Beck Depression Inventory (BDI) test.
Improvement of hearing loss - Fowler scoring | 36 months
  Improvement of the hearing loss in patients will be assessed using the pure-tone audiometry with Fowler scoring of hearing loss (%).

CONTACTS AND LOCATIONS:
Overall Officials: Michal Bar, Ass.Prof.,MD,PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD to other researchers has not been decided yet.

REFERENCES:
- [Background] Folmer RL, Carroll JR, Rahim A, Shi Y, Hal Martin W. Effects of repetitive transcranial magnetic stimulation (rTMS) on chronic tinnitus. Acta Otolaryngol Suppl. 2006 Dec;(556):96-101. doi: 10.1080/03655230600895465. PMID 17114152
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Kim BG, Kim DY, Kim SK, Kim JM, Baek SH, Moon IS. Comparison of the outcomes of repetitive transcranial magnetic stimulation to the ipsilateral and contralateral auditory cortex in unilateral tinnitus. Electromagn Biol Med. 2014 Sep;33(3):211-5. doi: 10.3109/15368378.2013.801353. Epub 2013 Jun 19. PMID 23781982
- [Background] Kleinjung T, Eichhammer P, Landgrebe M, Sand P, Hajak G, Steffens T, Strutz J, Langguth B. Combined temporal and prefrontal transcranial magnetic stimulation for tinnitus treatment: a pilot study. Otolaryngol Head Neck Surg. 2008 Apr;138(4):497-501. doi: 10.1016/j.otohns.2007.12.022. PMID 18359361
- [Background] Kreuzer PM, Landgrebe M, Schecklmann M, Poeppl TB, Vielsmeier V, Hajak G, Kleinjung T, Langguth B. Can Temporal Repetitive Transcranial Magnetic Stimulation be Enhanced by Targeting Affective Components of Tinnitus with Frontal rTMS? A Randomized Controlled Pilot Trial. Front Syst Neurosci. 2011 Nov 4;5:88. doi: 10.3389/fnsys.2011.00088. eCollection 2011. PMID 22069382
- [Background] De Ridder D, Song JJ, Vanneste S. Frontal cortex TMS for tinnitus. Brain Stimul. 2013 May;6(3):355-62. doi: 10.1016/j.brs.2012.07.002. Epub 2012 Jul 24. PMID 22853891
- [Background] Lehner A, Schecklmann M, Kreuzer PM, Poeppl TB, Rupprecht R, Langguth B. Comparing single-site with multisite rTMS for the treatment of chronic tinnitus - clinical effects and neuroscientific insights: study protocol for a randomized controlled trial. Trials. 2013 Aug 23;14:269. doi: 10.1186/1745-6215-14-269. PMID 23968498
- [Background] Lehner A, Schecklmann M, Poeppl TB, Kreuzer PM, Vielsmeier V, Rupprecht R, Landgrebe M, Langguth B. Multisite rTMS for the treatment of chronic tinnitus: stimulation of the cortical tinnitus network--a pilot study. Brain Topogr. 2013 Jul;26(3):501-10. doi: 10.1007/s10548-012-0268-4. Epub 2012 Dec 11. PMID 23229756
- [Background] Langguth B, Landgrebe M, Frank E, Schecklmann M, Sand PG, Vielsmeier V, Hajak G, Kleinjung T. Efficacy of different protocols of transcranial magnetic stimulation for the treatment of tinnitus: Pooled analysis of two randomized controlled studies. World J Biol Psychiatry. 2014 May;15(4):276-85. doi: 10.3109/15622975.2012.708438. Epub 2012 Aug 22. PMID 22909265
- [Background] Hoekstra CE, Versnel H, Neggers SF, Niesten ME, van Zanten GA. Bilateral low-frequency repetitive transcranial magnetic stimulation of the auditory cortex in tinnitus patients is not effective: a randomised controlled trial. Audiol Neurootol. 2013;18(6):362-73. doi: 10.1159/000354977. Epub 2013 Oct 19. PMID 24157459
- [Background] Engelhardt J, Dauman R, Arne P, Allard M, Dauman N, Branchard O, Perez P, Germain C, Caire F, Bonnard D, Cuny E. Effect of chronic cortical stimulation on chronic severe tinnitus: a prospective randomized double-blind cross-over trial and long-term follow up. Brain Stimul. 2014 Sep-Oct;7(5):694-700. doi: 10.1016/j.brs.2014.05.008. Epub 2014 Jun 4. PMID 25017670
- [Background] Plewnia C, Vonthein R, Wasserka B, Arfeller C, Naumann A, Schraven SP, Plontke SK. Treatment of chronic tinnitus with theta burst stimulation: a randomized controlled trial. Neurology. 2012 May 22;78(21):1628-34. doi: 10.1212/WNL.0b013e3182574ef9. Epub 2012 Apr 25. PMID 22539568
- [Background] Roland LT, Peelle JE, Kallogjeri D, Nicklaus J, Piccirillo JF. The effect of noninvasive brain stimulation on neural connectivity in Tinnitus: A randomized trial. Laryngoscope. 2016 May;126(5):1201-6. doi: 10.1002/lary.25650. Epub 2015 Sep 30. PMID 26422238
- [Background] Kleinjung T, Steffens T, Sand P, Murthum T, Hajak G, Strutz J, Langguth B, Eichhammer P. Which tinnitus patients benefit from transcranial magnetic stimulation? Otolaryngol Head Neck Surg. 2007 Oct;137(4):589-95. doi: 10.1016/j.otohns.2006.12.007. PMID 17903575
- [Background] Khedr EM, Rothwell JC, Ahmed MA, El-Atar A. Effect of daily repetitive transcranial magnetic stimulation for treatment of tinnitus: comparison of different stimulus frequencies. J Neurol Neurosurg Psychiatry. 2008 Feb;79(2):212-5. doi: 10.1136/jnnp.2007.127712. PMID 18202212
- [Background] Marcondes RA, Sanchez TG, Kii MA, Ono CR, Buchpiguel CA, Langguth B, Marcolin MA. Repetitive transcranial magnetic stimulation improve tinnitus in normal hearing patients: a double-blind controlled, clinical and neuroimaging outcome study. Eur J Neurol. 2010 Jan;17(1):38-44. doi: 10.1111/j.1468-1331.2009.02730.x. Epub 2009 Jul 9. PMID 19614962
- [Background] Frank G, Kleinjung T, Landgrebe M, Vielsmeier V, Steffenhagen C, Burger J, Frank E, Vollberg G, Hajak G, Langguth B. Left temporal low-frequency rTMS for the treatment of tinnitus: clinical predictors of treatment outcome--a retrospective study. Eur J Neurol. 2010 Jul;17(7):951-6. doi: 10.1111/j.1468-1331.2010.02956.x. Epub 2010 Feb 10. PMID 20158510
- [Background] Newman CW, Jacobson GP, Spitzer JB. Development of the Tinnitus Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1996 Feb;122(2):143-8. doi: 10.1001/archotol.1996.01890140029007. PMID 8630207
- See also: The American Academy of Audiology is the world's largest professional organization of, by, and for audiologists. — http://www.audiology.org